CLINICAL TRIAL: NCT05515029
Title: Prospective Pilot Study of the Clinical Efficacy and Safety of the Method for Preventing a Graft-versus-host Disease Through the Agency of Using the Combination of Post-transplantation Cyclophosphamide With Abatacept, Vedolizumab and Calcineurin Inhibitor at Children and Young Adults With Hemoblastosis After Hematopoietic Stem Cell Transplantation From an Unrelated or Haploidentic Donor
Brief Title: Preventing of GVHD With Post-transplantation Cyclophosphamide, Abatacept, Vedolizumab and Calcineurin Inhibitor at Patients With Hemoblastosis
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Federal Research Institute of Pediatric Hematology, Oncology and Immunology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCHPOI-2022-08
Record Dates: First submitted 2022-08-23; First posted 2022-08-25 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Acute Lymphoblastic Leukemia; Myeloblastic Leukemia; Biphenotypic Acute Leukemia; Malignant Lymphoma; Myelodysplastic Syndromes; Juvenile Myelomonocytic Leukemia
Keywords: Hematopoetic stem cell transplantation; posttransplant cyclophosphamide; vedolizumab; AML; ALL; children; graf versus host disease; adolescents
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelomonocytic, Acute; Leukemia, Biphenotypic, Acute; Lymphoma; Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Juvenile | interventions — Abatacept; vedolizumab; Calcineurin Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GVHD prevention: post-transplantation cyclophosphamide, abatacept, vedolizumab,calcineurin inhibitor (Experimental)
  Interventions: Combination Product: GVHD prevention: post-transplantation cyclophosphamide, abatacept, vedolizumab, calcineurin inhibitor

INTERVENTIONS:
Combination Product: GVHD prevention: post-transplantation cyclophosphamide, abatacept, vedolizumab, calcineurin inhibitor — Cyclophosphamide 100 mg/kg/course on the days +3, +4 Abatacept 10 mg/kg/day on the days +5, +14, +28, +45, +60, +90, +120 Vedolizumab 10 mg/kg/day, max. 300 mg on the days -1, +14, +28

SUMMARY:
GVHD prevention using a combination of post-transplantation cyclophosphamide in combination with abatacept, vedolizumab and calcineurin inhibitor in children and young adults with hematoloblastosis after myeloablative conditioning regimen with treosulfan/TBI, cyclophosphamide/etoposide, fludarabine after HSCT from matched unrelated and haploidentical donors

DETAILED DESCRIPTION:
Conditioning regimen:

Treosulfan 42 g/m2/course on the days -5, -4, -3 or total body irradiation 12 Gray/course on the days -8, -7, -6 Cyclophosphamide 50 mg/kg/course on the days -3, -2 or Etoposide 60 mg/kg on the days -6, -5 Fludarabine 150 mg/m2/course on the days -6, -5, -4, -3, -2

Prevention of GVHD:

Cyclophosphamide 100 mg/kg/course on the days +3, +4 Abatacept 10 mg/kg/day on the days +5, +14, +28, +45, +60, +90, +120 Vedolizumab 10 mg/kg/day, max. 300 mg on the days -1, +14, +28 Cyclosporine A or Tacrolimus 3 mg/kg/day from -1 to 120 (in case of high risk of relapse: patients with JMML, without of remission o positive MRD after HSCT)/180 days or Ruxolitinib (in case of intolerance to calcineurin inhibitors) 5m/day for patients <12 years old and 10 mg/day for patients >12 years old by scheme of CNI.

Donor selection criteria

In case of detection of two or more suitable donors, the choice is made in favor of:

* CMV Compliance
* Sex of donor and recipient
* medical and psychological suitability and desire of the donor
* Compatibility by blood type

Duration of therapy

* 120 days (for patients with high risk of recurrence: positive minimal residual disease before HSCT, non-remission status after HSCT, patients diagnosed with juvenile myelomonocytic leukemia)
* 180 days (for the rest) Time of observation
* follow up during 3 years after HSCT

Criteria for premature stopping of the study

1. The probability of developing acute GVHD II-IV is above 40%, of which III-IV - above 15%
2. The probability of 100-day transplant-associated mortality is higher than 20%. Goal Evaluation Date Intermediate analysis after 1 year from the beginning. The final analysis is scheduled to take place 100 days after the last patient is included.

Data Monitoring and Management

1. Plan of initial examination of the patient

After signing the informed consent and registration, the patient undergoes an examination in accordance with the standard plan of pre-transplantation examination and additional examinations, including:

* Confirmation of remission status, determination of MRD, chimerism according to the protocol 1. Monitoring of donor chimerism in patients with acute leukemia Point Days Lines

  1 +30 day general, CD34
* Only if a relapse of the disease is suspected, cm can be sent to study chimerism:

  * General
  * Chimerism in the sorted MRD fraction 2. Minimal residual disease (MRD) monitoring in patients with ALL +30, +100 days after HSCT - for all patients: MRD (immunophenotyping), Cytogenetics (if it presence)

    + 60, +180 days after HSCT - for patients with MRD + or refractory before HSCT: MRD (immunophenotyping), Cytogenetics (if it presence) 3. Minimal residual disease (MRD) monitoring in patients with AML

    +100 days after HSCT - for all patients: MRD (immunophenotyping), Cytogenetics (if it presence)

    + 30, +180 days after HSCT - for patients with MRD + or refractory before HSCT: MRD (immunophenotyping), Cytogenetics (if it presence)

    4. Biobanking (KM, blood)

In this protocol, in addition to routine post-transplantation monitoring, the following studies are carried out:

• Study of the subpopulation composition of peripheral blood lymphocytes: B-cells: CD19

T-cells:

CD3/4/8/ TCR/gd CD3/4/8/45RA/CCR7 (CD197) CD3/4/31/45RA CD4/25/127

NK-compartment:

CD3/CD56

TCR repertoire:

Analysis multiplicity: +30, +60, +100, +180, +360 day The amount of blood for analysis is 5 ml in a test tube with EDTA.

* Pathogen-specific immunoreconstitution research - ELISPOT method for evaluating the production of gamma-interferon by peripheral blood mononuclears after incubation with microbial antigens. The main antigens studied are (CMV pp65, EBV, Adenovirus (AdvHexon), BK virus) Multiplicity of analysis of recipients: +30, +60, +100, +180, +360. The amount of blood for analysis on +30 days is 10 ml, subsequently - 5 ml in a test tube with EDTA.
* Virological monitoring by PCR weekly:

Blood: CMV, EBV, ADV by PCR method Chair: ADV MONITORING by PCR is carried out up to 100 days after CGSC. The exception is patients with viremia, or receiving immunosuppressive therapy on day 100.

in case of suspected visceral lesion: cerebrospinal fluid / bal / stool / urine / biopsy / other material

* Biobanking Multiplicity: + 30, +60, +100, +180, +360 Blood in a test tube with EDTA, used 2. Toxicity monitoring:
* Diagnosis and therapy of acute GVHD Clinical diagnosis and staging of acute GVHD is carried out in accordance with standard criteria (Appendix No. 3).

When an isolated rash appears, a skin biopsy is mandatory. When a clinic of acute GVHD appears with damage to the upper and lower gastrointestinal tract (nausea, vomiting, enterocolitis), gastroscopy with a biopsy of the gastric mucosa and colonoscopy with a floor biopsy is reokended.

The biopsy material should also be sent for virological examination. Before starting therapy, a consultation is held with the head of the protocol / appointed expert.

• Criteria for prescribing systemic immunosuppressive therapy: Acute GVHD stage I - therapy is not carried out Acute GVHF stage II-IV - methylprednisolone 1-2 mg / kg / day IV The period for assessing the response to first-line therapy: 72 hours, 7 days, 14 days from the start of therapy.

• Criteria for prescribing second-line therapy: progression of manifestations of O.RTPH after 72 hours or no improvement after 7 days or incomplete resolution of clinical and laboratory manifestations after 14 days

• Diagnosis and therapy of chronic GVHD: Diagnosis and staging of chronic GVHD are performed in accordance with THE NIH criteria (Appendix No. 4). Due to the fact that the development of chronic GVHD is one of the main parameters for the evaluation of the study, the diagnosis and staging of chronic GVHD are performed prospectively, monthly from the day +100, using a structured examination in accordance with Appendix No. 2.

Therapy of chronic GVHD is carried out in accordance with the standard adopted in the clinic

ELIGIBILITY:
Inclusion Criteria:

Patients under the age of 21 years with following diseases:

* acute lymphoblastic,
* myeloblastic,
* biphenotypic,
* bilinear leukemia,
* malignant lymphoma,
* myelodysplastic syndrome,

Exclusion Criteria:

* Age over 21 years
* Patients with ALL outside clinical and hematological remission
* Clinical status:

  * Lansky/Karnowski index <70%
  * Heart function: left ventricular ejection fraction <40% according to ultrasound of the heart1
  * Kidney function: clearance of endogenous creatinine < 70 ml / min
  * Liver function: total bilirubin, ALT, AST, ALP > 2 norms
  * Lung function: lung capacity <50%, for children who cannot carry out of respiratory function - oxygen saturation during pulse oximetry <92%
* Uncontrolled viral, fungal or bacterial infection.
* Mental illness of the patient or caregivers, making it impossible to realize the essence of the study and compromising compliance with medical appointments and sanitary and hygienic regime 1 These patients may receive treatment according to the protocol, but the results will be evaluated separately

Ages: 1 Day to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 56 (Actual)
Dates: Start 2022-08-23 (Actual); Primary Completion 2024-08-15 (Estimated); Study Completion 2026-10-16 (Estimated)

PRIMARY OUTCOMES:
Estimate the probability of developing acute GVHD stage II-IV after HSCT | evaluation period is 120 days after HSCT
severe (3-5 degrees) side effects of conditioning | evaluation period is 30 days after HSCT

SECONDARY OUTCOMES:
event free survival | up to 100 days after HSCT
transplantation-associated mortality | up to 100 days after HSCT
relapse free survival | up to 100 days after HSCT
pathogen-specific immunoreconstitution | after HSCT up to 180 days
reactivation of CMV | after HSCT up to 180 days

CONTACTS AND LOCATIONS:
Locations (1):
- Dmitry Rogachev National Medical Research Center Of Pediatric Hematology, Oncology and Immunology, Moscow, Samory-Mashela,1, Russia